CLINICAL TRIAL: NCT03942380
Title: Cell-free Tumor DNAand HPV-DNA in Blood Samples From Newly Diagnosed Patients With Head and Neck Cancer
Brief Title: Cell-free Tumor DNA in Head and Neck Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christian von Buchwald (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other); Department of Otorhinolaryngology, Head and Neck Surgery and Audiology (Unknown)
Responsible Party: Sponsor-Investigator, Christian von Buchwald, Clinical Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1301261
Record Dates: First submitted 2019-04-15; First posted 2019-05-08 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms; Head and Neck Squamous Cell Carcinoma; Oropharynx Cancer; Oropharynx Neoplasm; Oropharynx Carcinoma; Oral Cavity Cancer; Oral Cancer; Oral Neoplasm; Larynx Cancer; Larynx Carcinoma; Larynx Neoplasm; Nasopharyngeal Carcinoma; Nasopharyngeal Cancer; Nasopharynx Neoplasm; Hypopharynx Cancer; Hypopharynx Neoplasm; Hypopharynx Carcinoma; Sinonasal Carcinoma; Thyroid Carcinoma; Thyroid Cancer; Thyroid Neoplasms; Salivary Gland Cancer; Salivary Gland Neoplasms; Salivary Gland Carcinoma; Sinonasal Cancer; Sinonasal Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Mouth Neoplasms; Laryngeal Neoplasms; Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Hypopharyngeal Neoplasms; Thyroid Neoplasms; Salivary Gland Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cell-free tumor DNA (Other): The aim is to differentiate between patients with head and neck cancer from those without based on a blood sample.
  Interventions: Diagnostic Test: Liquid biopsy
- Identifying recurrence (Other): The aim is to identify recurrence through serial monitoring patients with blood samples.
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — The intervention is a liquid biopsy as a blood sample taken in a peripheral vein. The blood samples are analyzed for cell free DNA, RNA and HPV-DNA

SUMMARY:
This study investigates if head and neck squamous cell carcinoma can be tracked with cell-free tumor DNA, RNA or HPV-DNA, in blood samples from patients referred with suspicion of cancer, and if it can be used in detecting recurrence in patients already diagnosed and treated for head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Suspicion of head and neck cancer

Exclusion Criteria:

* Diagnosed with cancer within the last 3 years ( apart from basal cell carcinoma)
* Diagnosed with an inflammatory or haematological disease after the age of 18
* Received chemotherapy or immunosuppressive treatment within the last 3 years
* Underwent a FNA ( fine-needle aspiration biopsy) or a biopsy from the head and neck region within 1 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of head and neck cancer detected with a blood sample | 0 months
  The primary outcome is to measure the percentage of head and neck squamous cell carcinomas that can be detected using a liquid biopsy (blood sample)
Percentage of head and neck cancer recurrence detected with a blood sample | 36 months
  The primary outcome is to measure the percentage of recurrence in head and neck cancer patients through serial monitoring with liquid biopsies (blood sample)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Von Buchwald, MD, DMSc, Principal Investigator — Department of Otorhinolaryngology, Head and Neck Surgery and Audiology
Locations (1):
- University Hospital of Copenhagen, Rigshospitalet, Copenhagen, Capital Region, Denmark